CLINICAL TRIAL: NCT03429985
Title: Fathers Raising Responsible Men (FRRM): Addressing Sexual Health to Reduce Teen Pregnancy
Brief Title: Fathers Raising Responsible Men (FRRM): Addressing Sexual Health
Acronym: FRRM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: In response to the COVID pandemic, and in accordance with local and university public health restrictions, our team suspended the study. This disrupted all planned follow-up activities. With funder approval, we pivoted our project to a non-RCT design
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRO00108880
Record Dates: First submitted 2017-09-15; First posted 2018-02-12 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Behavior and Behavior Mechanisms
Keywords: Sexual and Reproductive Health; Parent-based Intervention; Sexual Risk Behavior; Adolescent Males; Father-Son Intervention; Life Opportunities
MeSH Terms: conditions — Behavior; Coitus

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FRRM Intervention (Experimental): The experimental arm will receive the FRRM intervention.
  Interventions: Behavioral: FRRM Intervention
- Control (No Intervention): The control arm will not receive the FRRM intervention.

INTERVENTIONS:
Behavioral: FRRM Intervention — Fathers Raising Responsible Men (FRRM) is designed to facilitate important paternal parenting behaviors that influence adolescent decision-making. FRRM incorporates a novel, theoretically-based intervention highlighting the important and influential role that fathers have on the development and life trajectories of adolescent males.
  Other Names: FRRM
  Arms: FRRM Intervention

SUMMARY:
While existing teen pregnancy prevention efforts have contributed to significant declines in the overall U.S. teen pregnancy rate, teen pregnancy prevention programs specifically targeting adolescent males are limited and sorely needed. The primary aim of the proposed research is to further develop, evaluate, and disseminate a teen pregnancy prevention program specifically designed for adolescent males to enhance the current scientific evidence and intervention options available for broad public health implementation. The proposed intervention Fathers Raising Responsible Men (FRRM) focuses on the adolescent male component of teen pregnancy by identifying and addressing adolescent risk and paternal protective behaviors specific to adolescent males that have not been fully addressed in previous prevention efforts. This study strives to reduce adolescent male sexual risk behavior through targeting African American and Latino adolescent males aged 15-19 and their fathers residing in the South Bronx, specifically Mott Haven and surrounding areas in three phases. Phase I is a pilot study consisting of eight dyads (fathers and sons) to test and refine the intervention and technical and training assistance needs. Phase II is the Randomized Control Trial (RCT) comprised of two cohorts (a total of 500 father-son dyads) to rigorously evaluate the intervention. During the final 6 months of the project, qualitative interviews with 30 father-son dyads will be conducted to triangulate the quantitative RCT results with participant experiences of FRRM. Finally, in Phase III the intervention will be refined and the intervention materials will be available to the general public, while findings will be widely disseminated. These three phases allow for the successful implementation and evaluation of FRRM in conjunction with the refinement and provision of all training and technical assistance necessary for the intervention. If successful, the proposed project will further develop the current scientific evidence and intervention options targeted specifically to the teen pregnancy prevention needs of African American and Latino adolescent males.

DETAILED DESCRIPTION:
FRRM is a male-focused intervention designed to reduce adolescent male sexual risk behavior through supporting father-son communication about sex and condoms, as well as improve future life trajectories. The goals of the program are to reduce the number of unprotected sex acts among adolescents through (1) improved knowledge about correct and consistent condom use, (2) increased sexual transmitted infection (STI) testing, and (3) increased utilization of sexual and reproductive health services. Additionally, the program aims to improve adolescent life opportunities through (1) improved perception of life trajectories; and (2) increased utilization of academic and job training services within the community.

The RCT consists of two cohorts. The first cohort (n=200 father-son dyads) will receive (1) two 60 to 90 minute intervention sessions delivered to the father by project staff. Intervention sessions should happen within the first month following the baseline interview. The first intervention session focuses on motivating fathers to communicate with their sons about sex and condom use, and the second session provides fathers with the skills and knowledge necessary to teach their sons about correct condom use. In addition, fathers receive guidance on effective adolescent monitoring and supervision and strengthening their relationship quality with their adolescent son.

The second cohort (n=300 father-son dyads) will receive (1) two 60 to 90 minute intervention sessions delivered to the father by project staff with content identical to the interventions given to cohort one; and 2) one 60 to 90 minute intervention session delivered to the father-son dyad by project staff regarding adolescent life opportunities. In the third intervention session, the father coach provides father-son dyads with specific guidance and helpful resources for on-going and positive interactions between fathers and sons. Additionally, this session highlights specific academic and job training resources within the community that fathers and sons can access to better address adolescent sexual and reproductive health, overall wellbeing, and future goals/aspirations.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the study, adolescent sons must:

1. be 15 to 19 year old male,
2. identify as either African American or Latino,
3. reside in one of the four target neighborhoods in the South Bronx, and
4. not be a teen father, married, or co-habitating with his partner.

Eligible fathers must:

1. be the primary caregiver who is male of the target son (this can include biological fathers, grandfathers, and uncles).
2. Reside in Mott Haven or surrounding areas of the South Bronx or other parts of New York City; able to meet with son at son's primary residence or mutually agreed-upon location.

Exclusion Criteria:

Both fathers and sons must not be participating in any other teen pregnancy prevention program at the start of the study.

Ages: 15 Years to 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 382 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Number of Unprotected Sex Acts Among Adolescent Males | Delayed follow up (9 months)
  Defined as number of sex acts without using a contraceptive method

SECONDARY OUTCOMES:
Adolescent Consistency of Condom Use: As Measured by the Condom Use Among Hispanics Scale | Delayed follow up (9 months)
  Defined as frequency of adolescent condom use during sex acts
Adolescent Frequency of Sex Acts | Delayed follow up (9 months)
  Defined as number of sex acts within a time period
Adolescent Knowledge of Correct Condom Use: As Measured by the Condom Use Among Hispanics Scale | Delayed follow up (9 months)
  Defined as adolescent knowledge of the correct steps of using a condom, with higher scores indicating greater knowledge of the five steps of condom use.
Adolescent Attendance at Sexual and Reproductive Health Service | Delayed follow up (9 months)
  Defined as adolescent report of having attended a sexual and reproductive health visit
Adolescent HIV Testing Results | Delayed follow up (9 months)
  Defined as the prevalence of HIV at follow-up
Adolescent Gonorrhea Testing Results | Delayed follow up (9 months)
  Defined as the prevalence of gonorrhea at follow-up
Adolescent Chlamydia Testing Results | Delayed follow up (9 months)
  Defined as the prevalence of chlamydia at follow-up
Adolescent Attendance at Job Training Services | Delayed follow up (9 months)
  Defined as adolescent report of having attended a job training services visit
Adolescent Attendance at Educational Support Services | Delayed follow up (9 months)
  Defined as adolescent report of having attended an educational support services visit
Adolescent Attendance at Wraparound Services | Delayed follow up (9 months)
  Defined as adolescent report of having attended a wraparound services visit
Adolescent Perception of Future Academic and Career Success: As Measured by the Perceived Life Chances Scale | Delayed follow up (9 months)
  Defined as adolescent report of their perceived likelihood of achieving future goals and aspirations, with higher scores indicating greater perceived likelihood of achieving long-term goals.
Number of Unprotected Sex Acts Among Adolescent Males | Immediate follow up (3 months)
  Defined as number of sex acts without using a contraceptive method
Adolescent Consistency of Condom Use: As Measured by the Condom Use Among Hispanics Scale | Immediate follow up (3 months)
  Defined as the proportion of total sex acts where a condom was used, with higher scores indicating a greater percentage of condom use.
Adolescent Frequency of Sex Acts | Immediate follow up (3 months)
  Defined as number of sex acts within a time period
Adolescent Knowledge of Correct Condom Use: As Measured by the Condom Use Among Hispanics Scale | Immediate follow up (3 months)
  Defined as adolescent knowledge of the correct steps of using a condom, with higher scores indicating greater knowledge of the five steps of condom use.
Adolescent Attendance at Sexual and Reproductive Health Services | Immediate follow up (3 months)
  Defined as adolescent report of having attended a sexual and reproductive health visit
Adolescent HIV Testing Results | Immediate follow up (3 months)
  Defined as the prevalence of HIV at follow-up
Adolescent Gonorrhea Testing Results | Immediate follow up (3 months)
  Defined as the prevalence of gonorrhea at follow-up
Adolescent Chlamydia Testing Results | Immediate follow up (3 months)
  Defined as the prevalence of chlamydia at follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University School of Nursing, New York, New York, United States